CLINICAL TRIAL: NCT05937880
Title: Leflunomide for Refractory Skin Henoch-Schonlein Purpura in Children
Brief Title: Leflunomide for Henoch-Schonlein Purpura
Acronym: Lef for HSP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Weiping Tan, Professor, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-KY-002
Record Dates: First submitted 2023-06-25; First posted 2023-07-10 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Henoch-Schonlein Purpura
Keywords: Leflunomide; Henoch-Schonlein Purpura; Children; Efficacy
MeSH Terms: conditions — IgA Vasculitis | interventions — Leflunomide

STUDY DESIGN:
Intervention Model Description: Refractory skin Henoch-Schonlein Purpura
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Administration of Leflunomide in refractory skin Henoch-Schonlein purpura (Experimental): Rashes are dense and large in area, often treated with antibiotics, antihistamines, calcium supplements, and glucocorticoids (2 mg/kg/d) for 5 days. The rash does not subside or new rash still appears, and it frequently repeats more than 3 times during hospitalization.
  Interventions: Drug: Leflunomide

INTERVENTIONS:
Drug: Leflunomide — When patients appeared with rashes and treated with antibiotics, antihistamines, calcium supplements, and glucocorticoids (2 mg/kg/d) for 5 days. The rashes do not subside or fresh rash still appears, and it frequently repeats more than 3 times during hospitalization. Leflunomide would be administered

SUMMARY:
This study conducted a prospective, multicenter, one-arm clinical trial on the combination of leflunomide and steroid therapy for refractory skin Henoch-Schonlein Purpura in children on the basis of ethical principles. A one-year follow-up was conducted to evaluate the changes in the main indicators (frequency of rash recurrence) and secondary indicators (proportion of kidney damage, proportion of joint involvement, T lymphocyte subpopulations, and inflammatory factors) before and after treatment, Exploring the safety and effectiveness of leflunomide in the treatment of refractory skin type HSP in children, it is expected that leflunomide combined with conventional treatment can improve the remission rate of HSP children's skin purpura and reduce HSP recurrence. The research results are expected to bring new treatment methods and strategies for this group of patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age ranges from 1 to 18 years old;
2. Patients meet the HSP diagnostic criteria;
3. Refractory skin type HSP: Rashes are dense and large in area, often treated with antibiotics, antihistamines, calcium supplements, and glucocorticoids (2 mg/kg/d) for 5 days. The rash does not subside or fresh rash still appears, and frequently repeated more than 3 times during hospitalization.
4. Parents or guardians agree to treatment and sign a written informed consent form.

Exclusion Criteria:

1. Individuals who are allergic to leflunomide;
2. Concomitant severe underlying diseases (such as systemic malignancy, heart failure, liver and kidney failure, immune deficiency, severe infectious diseases, organ transplant surgery, or other current indications for emergency surgery);
3. Patients with other digestive system diseases;
4. Those who have previously used flumiphene in clinical trials;
5. Excluding purpura caused by drugs, infectious factors, and other autoimmune diseases.
6. Other situations where the researcher deems it inappropriate to participate in the study.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Rash frequency | 12 months
  Rash frequency in a months

CONTACTS AND LOCATIONS:
Overall Officials: Weiping Tan, PhD, Study Chair — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No